CLINICAL TRIAL: NCT03294746
Title: Qualification of Imaging Methods to Assess Cancer Drug Induced Interstitial Lung Disease (ImageILD)
Brief Title: Imaging Biomarker in Cancer Drug Induced ILD
Acronym: ImageILD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EORTC-1658-IG
Record Dates: First submitted 2017-09-01; First posted 2017-09-27 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Drug Induced Interstitial Lung Disease (DIILD) Cancer Patients
Keywords: Drug induced interstitial lung disease (DIILD)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical evaluations and Thoracic CT scan scoring of DIILD (Other)
  Interventions: Other: Clinical evaluations; Other: Thoracic CT

INTERVENTIONS:
Other: Clinical evaluations — At study entry , 6 weeks and 6 months, enrolled patients will undergo pulmonary physiology tests, assessment of respiratory symptoms, respiratory examination, pulse oximetry, blood draws, respiratory and quality of life assessment. Data from bronchoscopy assessments will be collected, if this has been performed as part of routine care.
Other: Thoracic CT — At study entry, patients will undergo thoracic CT before treatment adaptation, unless a study-quality scan* has already been performed . Thoracic CT will be repeated at 6 weeks. All images will be centrally reviewed for radiology scoring.

SUMMARY:
Drug induced interstitial lung disease (DIILD) is caused by iatrogenic injury to the lung parenchyma and can be caused by over four hundred different drugs in humans. Diagnosing DIILD is a challenge for clinicians and radiologists as a positive diagnosis depends on exclusion of other causes including respiratory infection, occupational, recreational, and environmental exposures, specific respiratory disorders, and systemic diseases.

The aim of this study is to qualify an objective CT scoring system for DIILD assessment. In addition, the quantitative information obtained from CT scans with densitometry and texture analysis will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* World health organization (WHO) performance status 0-2
* Life expectancy > 6 months
* Proven cancer diagnosis in a patient actively undergoing anti-cancer therapy
* New onset symptoms (e.g. cough, fever, dyspnoea, and hypoxia) at any time during or within 4 weeks of the last dose of anti-cancer treatment
* New onset radiological (CXR or CT) abnormalities within the lungs at any time during or within 4 weeks of the last dose of anti-cancer treatment (e.g. diffuse lung changes, infiltrative opacification in the periphery of the lung or ground glass changes) with a locally reviewed diagnosis of DIILD as the most likely explanation for the radiological abnormalities.
* Treatment for DIILD planned (e.g. drug withdrawal, interruption +/- supportive therapy including corticosteroids, oxygen, bronchodilators etc.). Concomitant treatment with antibiotics, anticoagulants etc. is permitted pending results of investigations for differential diagnoses.
* Able to undergo pulmonary function tests (at a minimum spirometry and gas transfer (DLCO))
* Patients enrolled on other anti-cancer investigational trials are permitted at investigator discretion
* Informed written consent obtained according to national/local regulations
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 14 days before study registration

Exclusion Criteria:

* Clinically suspected or confirmed radiological features of any malignancy involving the lungs at the time of study registration
* Claustrophobia, or inability to undergo non-contrast CT examination
* Known or suspected non-drug related ILD (e.g. lung abnormalities due to other causes such as occupational exposure)
* Previous extensive thoracic surgery (e.g. lobectomy)
* Clinical, radiological or microbiological evidence of active lower respiratory tract infection
* Currently active, clinically significant heart disease, such as uncontrolled class 3 or 4 congestive heart failure defined by the New York Heart Association Functional Classification
* Any medical, psychological, sociological or geographical condition that could affect participation in the study and compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient between semi-quantitative CT score and FVC (forced vital capacity) | analyses will be performed 3.5 years after First Patient In
  The primary objective of the study is to qualify an objective semi-quantitative CT scoring system looking at the correlation between the change in the semi-quantitative CT score at 6 weeks relative to baseline (DIILD diagnosis) against the change in Forced vital capacity (FVC) at 6 weeks relative to baseline (DIILD diagnosis). The semi-quantitative CT score will be calculated based on CT features: 1)ground-glass opacity 2) reticular/septal lines 3) honeycombing 4) nodular opacity 5) consolidation.

SECONDARY OUTCOMES:
Correlation coefficient between the semi-quantitative CT score with the other pulmonary physiology measurements (DLCO and 6WMT) and patient reported outcome (respiratory and quality of life). | analyses will be performed 3.5 years after First Patient In
To evaluate the predictive value of change in the semi-quantitative CT score. | analyses will be performed 3.5 years after First Patient In
  To evaluate the predictive value of change in the semi-quantitative CT score at 6 weeks relative to baseline (DIILD diagnosis) against change in pulmonary physiology measurements and patient reported outcome (respiratory and quality of life) at 6 months relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Linton, Principal Investigator — The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All publications must comply with the terms specified in the EORTC Policy 009 "Release of Results and Publication Policy".